CLINICAL TRIAL: NCT01161875
Title: Study of the Benefit of the NAVA Mode Versus PSV Mode on Patient Ventilator Asynchrony During Non Invasive Ventilation With Helmet
Brief Title: Impact of Neurally Adjusted Ventilator Assist (NAVA) Mode on Patient Ventilator Asynchrony Using Helmet
Acronym: NAVAHELMET
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Professor Thomas SIMILOWSKI, Groupe Hospitalier Pitie Salpetriere
Other Study IDs: Nava Helmet #1
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2009-11

CONDITIONS: Non-Invasive Positive-Pressure Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Neurally Adjusted Ventilatory Assistance — In ICU following abdominal aortic surgery, in extubated patient, non-invasive ventilation was performed as follows:
  * facial mask with non-invasive pressure support ventilation mode to define settings for helmet ventilation
  * helmet use with non-invasive pressure support ventilation mode to define adequate settings
  * helmet use with neurally adjusted ventilatory assist mode, based on previous settings

SUMMARY:
Non invasive ventilation has been proposed to reduce the incidence of ventilatory dysfunction following abdominal aortic surgery. However, the nasogastric tube reduces the airtightness of the facial mask used to perform non invasive ventilation and induces air leaks. The use of a helmet reduces air leaks, thus seems adequate to ensure patient-ventilator interface. However, the high dead space related to helmet volume is responsible for asynchrony between patient demand and ventilatory support delivery. The investigators hypothesized driving the ventilator based on a neural signal (diaphragm electrical activity) would reduce patient-ventilator asynchronies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with increased risk of postoperative ventilatory dysfunction following abdominal aortic surgery

Exclusion Criteria:

* Contra-indication to non-invasive ventilation pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative period
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Triggering delay | Every inspiration, for 10 minutes
  Duration between the onset of neural inspiration and the onset of insufflation

SECONDARY OUTCOMES:
Cycling off delay | Every inspiration, for 10 minutes
  Delay between the end of neural inspiration and the end of insufflation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Similowski, MD, PhD, Study Director — Groupe Hospitalier Pitie-Salpetriere; Mathieu RAUX, MD, PhD, Principal Investigator — Groupe Hospitalier Pitie-Salpetriere
Locations (1):
- Groupe Hospitalier Pitie Salpetriere, Department of Anesthesiology and Critical Care, Paris, France